CLINICAL TRIAL: NCT06137287
Title: BOTOX VISTA® (onabotulinumtoxinA) for Masseter Muscle Prominence: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: A Study to Assess Adverse Events and Change of Masseter Muscle Prominence Using BOTOX Injections in Adult Participants
Acronym: MMP Japan 080
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M22-080
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Masseter Muscle Prominence
Keywords: Masseter Muscle Prominence; OnabotulinumtoxinA; BOTOX VISTA; BOTOX
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (Experimental): In Period 1, participant will receive 6 injections of BOTOX VISTA Dose A on Day 1. In Period 2, participants who meet the retreatment criteria will receive 6 injections of BOTOX VISTA Dose A on either Day 180, 210, 240, or 270.
  Interventions: Drug: BOTOX
- Group 2 (Experimental): In Period 1, participant will receive 6 injections of BOTOX VISTA Dose B on Day 1. In Period 2, participants who meet the retreatment criteria will receive 6 injections of BOTOX VISTA Dose B on either Day 180, 210, 240, or 270.
  Interventions: Drug: BOTOX
- Group 3 (Experimental): In Period 1, participant will receive 6 injections of BOTOX VISTA placebo on Day 1. In Period 2, participants who meet the retreatment criteria will receive 6 injections of BOTOX VISTA Dose A on either Day 180, 210, 240, or 270.
  Interventions: Drug: BOTOX; Drug: Placebo for BOTOX
- Group 4 (Experimental): In Period 1, participant will receive 6 injections of BOTOX VISTA placebo on Day 1. In Period 2, participants who meet the retreatment criteria will receive 6 injections of BOTOX VISTA Dose B on either Day 180, 210, 240, or 270.
  Interventions: Drug: BOTOX; Drug: Placebo for BOTOX

INTERVENTIONS:
Drug: BOTOX — Intramuscular Injection
  Other Names: BOTOX VISTA; OnabotulinumtoxinA
Drug: Placebo for BOTOX — Intramuscular Injection
  Arms: Group 3; Group 4

SUMMARY:
The masseter muscle is one of the muscles in the lower face used for chewing. Prominence of the masseter muscle can appear as a widened and square lower face shape, which is an aesthetic concern for individuals who prefer a narrower and more ovoid lower face shape. Treatments are available for masseter muscle prominence (MMP), but researchers are looking for new non-surgical treatments. This study will assess adverse events and effectiveness of BOTOX in adult participants with MMP.

BOTOX is being investigated for the treatment of MMP. Participants are placed in 1 of 4 groups, called treatment arms. Each group receives a different treatment. There is 1 in 5 chance that participants will be assigned to placebo. Around 250 adult participants with MMP will be enrolled in the study at approximately 20 sites in Japan.

Participants will receive either BOTOX or Placebo administered as 6 intramuscular injections to each masseter muscle on Day 1. Participants who are eligible for retreatment will be given BOTOX on either Day 180, 210, 240, or 270 and will be followed until approximately Day 360.

There may be a higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, facial photography, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Adult Japanese individuals.
* Participant with marked or very marked masseter muscle prominence (MMP).

Exclusion Criteria:

* Asymmetry of left and right sides of the face that could prevent identical Masseter Muscle Prominence Scale (MMPS) or MMPS-P grading on both sides of the face, as determined by the investigator.
* History of permanent soft tissue fillers in the jawline.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 259 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve >= 2-Grade Improvement on Investigator-Rated Masseter Muscle Prominence Scale (MMPS) | Baseline to Day 90
  The MMPS is a photonumeric scale encompassing visual inspection of the masseter muscles as performed by the investigator, where the masseter muscle prominence (MMP) is rated at rest, by separately evaluating the left and right side of the participant's face. The evaluation is on a 5-grade scale where 1 = the masseter muscle prominence is minimal and 5 = the masseter muscle prominence is very marked.
Number of Participants with Adverse Events (AEs) | Up to approximately 12 months
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment

SECONDARY OUTCOMES:
Change from Baseline in Lower Facial Volume (cm^3) | Baseline to Day 90
  Photographic technologies developed to provide 3D quantitative analysis of facial morphology include image subtraction technique, moire topography, liquid crystal scanning, light luminance scanning, laser scanning, stereo-lithography, and passive stereophotogrammetry, which all measure change to the lower facial contour.
Change from Baseline in Lower Facial Width (mm) | Baseline to Day 90
  Photographic technologies developed to provide 3D quantitative analysis of facial morphology include image subtraction technique, moire topography, liquid crystal scanning, light luminance scanning, laser scanning, stereo-lithography, and passive stereophotogrammetry, which all measure change to the lower facial contour.
Percentage of Participants with Responses of Very Satisfied or Satisfied on the Lower Facial Shape Questionnaire - Treatment Satisfaction (LFSQ-TXSAT) Follow-Up Version | Day 90
  The LFSQ-TXSAT at follow-up measures the participant's satisfaction with the effect of treatment on the appearance of their lower face based on a 5-point scale where 2 = very satisfied and -2 = very dissatisfied.
Responses of Not at All Bothered or A Little Bothered on the Bother Impact Assessment for Masseter Muscle Prominence (BIA-MMP) (for Subjects Somewhat Bothered, A Lot Bothered, or Extremely Bothered at Baseline) | Day 90
  The BIA-MMP is a single item evaluation of how bothered the participant is by the appearance of their lower face using a 5-point scale where 0 = not at all bothered and 4 = extremely bothered.
Percentage of Participants who Achieve >= 2-Grade Improvement on Masseter Muscle Prominence Scale - Participant (MMPS-P) | Baseline to Day 90
  The MMPS-P is a patient reported outcomes (PRO) measure with an accompanying photo guide used to assess MMP severity from the participant perspective using a 5-grade scale where 1 = the muscle is not at all noticeable and 5 = the muscle is extremely noticeable.
Change from Baseline in Lower Facial Shape Questionnaire - Impact Assessment (LFSQ-IA) Summary Score | Baseline to Day 90
  The LFSQ-IA is a 6-item assessment that measures psychosocial impact of the appearance of the lower face using a 5-point scale where 0 = not at all and 4 = extremely.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- Japan (18):
  - Jyosui Dermatology Clinic /ID# 254300, Fukuoka, Fukuoka
  - Kotoni Tower Skin And Cosmetic Surgery Clinic /ID# 260668, Sapporo, Hokkaido
  - Tokai University Hospital /ID# 254204, Isehara, Kanagawa
  - Yoshikawa Skin Ecru Clinic /ID# 256505, Kyoto, Kyoto
  - Touyama Plastic Surgery Clinic /ID# 254831, Naha, Okinawa
  - Dermatology and Ophthalmology Kume Clinic /ID# 254632, Sakai-shi, Osaka
  - Skin Clinic Fujieda /ID# 254214, Fujieda-shi, Shizuoka
  - Tokyo Center Clinic /ID# 254775, Chuo-ku, Tokyo
  - Tokyo Asbo Clinic /ID# 257728, Chuo-ku, Tokyo
  - Ginza Skin Clinic /ID# 254666, Chuo-ku, Tokyo
  - Jiyugaoka Clinic /ID# 256666, Meguro-ku, Tokyo
  - Azabu beauty clinic /ID# 254519, Minato, Tokyo
  - Roppongi Imaizumi Skin Clinic /ID# 254573, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 255369, Minato-ku, Tokyo
  - Greenwood Skin Clinic Tachikawa /ID# 254830, Tachikawa-shi, Tokyo
  - Ikebukuronishiguchi Fukurou Dermatology Clinic /ID# 254639, Toshima-ku, Tokyo
  - Jun Clinic /Id# 254870, Nagano
  - Chiharu Dermatology Clinic Urawa /ID# 254778, Saitama

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-080